CLINICAL TRIAL: NCT02749461
Title: Validation of the Bernese Pain Scale for Neonates With Consideration for Contextual Factors
Brief Title: Validation of the Bernese Pain Scale for Neonates
Acronym: BERN-PAIN
Status: Completed | Type: Observational
Sponsor: Bern University of Applied Sciences (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other); University of Zurich (Other); University Children's Hospital Basel (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Eva Cignacco, Prof. Dr., Bern University of Applied Sciences
Other Study IDs: SNF 320030_159573
Record Dates: First submitted 2016-04-12; First posted 2016-04-25 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Pain Assessment
Keywords: preterm infants; pain; assessment; contextual factors; diagnostic accuracy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: heel stick — Consecutive routine blood sampling heel sticks

SUMMARY:
The aims of this validation study are the testing of the Bernese Pain Scale for Neonates' (BPSN) psychometric properties. The variability of pain reactions related to behavioral and physiological patterns across time will also be examined. Furthermore, the influence of contextual factors on the variability of pain reactions across gestational age groups will be explored. The results will be used for modifications of the BPSN to account for contextual factors in future clinical pain assessment in neonates.

DETAILED DESCRIPTION:
Preterm birth rates are rising worldwide, including in Europe. In 2014, Switzerland's rate of premature births reached 7.2%. Still, while significant progress in neonatal care has increased the long-term survival of preterm infants, other long-term outcomes remain problematic. As a result, affected infants commonly undergo exceedingly high numbers of painful procedures on a daily basis. For many, these treatment interventions take place at a crucial period in the development of the nociceptive and central nervous systems, i.e., at a developmental stage when repeated painful stimulus may induce both structural and functional reorganization of the nervous system and an altered pain response.

As infants are unable to communicate verbally, clinical pain assessment in neonates, particularly those delivered preterm, is highly challenging. Therefore, pain responses have to be observed according to physiological and behavioral indicators which might vary across preterm infants depending on their physiological and neurological development stages.

The Bernese Pain Scale for Neonates (BPSN) is a multidimensional pain assessment tool which is already widely used in clinical settings in the German speaking areas of Europe. Recent findings suggest that pain reaction is influenced by more than noxious stimulation alone: it is assumed that contextual factors, e.g., gestational age (GA) or gender, might also impact pain reactivity.

The aims of this validation study are:

* to undertake the psychometric testing of the BPSN regarding its concurrent validity with the Premature Infant Pain Profile-Revised (PIPP-R), construct validity, interrater and intrarater reliability, specificity and sensitivity;
* to examine the variability of pain reactions related to behavioural and physiological patterns across time;
* to assess the influence of contextual factors on the variability of pain reactions across GA groups; and
* to examine the relationship between behavioural and physiological indicators across time.

This multisite psychometric measurement study of the BPSN will use repeated measures design. The study will take place in three tertiary care hospitals (Bern, Zurich and Basel) in Switzerland. To examine the impact of GA on pain reaction and its variability, the infants will be stratified into six GA groups ranging from 24 0/7 to 42 0/7. Among preterm infants with GAs up to 36 6/7 weeks, five consecutive heel sticks within the first 14 days of life will be documented. Among healthy-term infants two heel sticks within the first days after birth will be documented. For each heel stick, measurements will be recorded for each of three phases: baseline, heel stick, and recovery. All phases will be videotaped and the child's pain reaction later rated according to the BPSN by five independent raters blinded to the measurement phase. Individual contextual factors of interest for this study are documented in a standardised way in all three participating Neonatal Intensive Care Units (NICUs), and can be extracted from patient charts.

This diagnostic study is intended to validate the BPSN with consideration for contextual factors influencing neonatal pain responses. Understanding and embedding the influences of contextual factors into a final version of the BPSN-Context will help clinicians more accurately assess pain in the clinical setting, and will eventually help them minimize the pain endured by neonates, particularly preterm neonates in NICUs. For preterm infants requiring intensive care, adequate and efficient pain management is an important factor in later motor and cognitive development. The investigators hope this study will contribute to the prevention of negative long-term outcomes in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born between 24 0/7 and 36 6/7 weeks of gestation will be included if they are expected to undergo 5 routine heel capillary blood samples during the first 14 days of life; if they are ventilated or not ventilated; and if their parents give informed consent.
* Term infants born between 37 0/7 and 42 0/7 weeks of gestation will be included if they are expected to have at least 2 routine heel capillary blood samples during the first days of life and if their parents give informed consent.

Exclusion Criteria:

* Grade III oder IV intraventricular haemorrhaging
* Severe life-threatening malformation or suffer from any condition involving partial or total loss of sensitivity
* pHa < 7.15 (umbilical cord)
* Surgery for any reason
* Congenital malformation affecting brain circulation and cardiovascular system

Ages: 24 Weeks to 41 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study includes preterm infants born between 24 0/7 and 36 6/7 weeks of gestation and term infants born between 37 0/7 and 42 0/7 weeks of gestation if they are hospitalised in a NICU in the University Hospitals in Basel, Bern and Zurich (Switzerland).
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2015-11; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in pain response across time | 2-5 timepoints within the first 14 days of life
  Change and variability of pain response across different time points will be measured with the BPSN

SECONDARY OUTCOMES:
Influence of individual contextual factors on pain response across time | 2-5 within the first 14 days of life
  Time points of contextual factors documentation are determined by the clinical need for routine heel stick procedures within the first 14 days of life. These time points are not fixed before hand but are based on ongoing clinical judgement during the first 14 days of life. For each clinically determined time point for a heel stick appropriate contextual factors being relevant the day of the determined heel stick date will be extracted from patient chart.
Psychometric testing of the BPSN | 2-5 timepoints within the first 14 days of life
  Psychometric testing will be done across all the five time points for baseline, heel stick and recovery phases

CONTACTS AND LOCATIONS:
Overall Officials: Eva Cignacco, Prof. Dr., Principal Investigator — Bern University of Applied Sciences
Locations (4):
- Lawrence S. Bloomberg Faculty of Nursing and Faculties of Medicine and Dentistry, University of Toronto, Toronto, Canada
- Switzerland (3):
  - Department of Neonatology, University Children's Hospital of Basel (UKBB), Basel
  - Neonatology, Children's Hospital, University Hospital of Bern, Bern
  - Neonatology, University Hospital of Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schenk K, Stoffel L, Burgin R, Stevens B, Bassler D, Schulzke S, Nelle M, Cignacco E. The influence of gestational age in the psychometric testing of the Bernese Pain Scale for Neonates. BMC Pediatr. 2019 Jan 15;19(1):20. doi: 10.1186/s12887-018-1380-8. PMID 30646872
- [Derived] Cignacco E, Schenk K, Stevens B, Stoffel L, Bassler D, Schulzke S, Nelle M. Individual contextual factors in the validation of the Bernese pain scale for neonates: protocol for a prospective observational study. BMC Pediatr. 2017 Jul 19;17(1):171. doi: 10.1186/s12887-017-0914-9. PMID 28724434
- See also: Swiss National Science Foundation (SNSF), grant database — http://p3.snf.ch/project-159573